CLINICAL TRIAL: NCT02943200
Title: The Prevalence of Malocclusion Development in a Group of Egyptian Children With Digit Sucking Aged 3 to 6 Years: A Cross Sectional Study
Brief Title: The Prevalence of Malocclusion Development in a Group of Egyptian Children With Digit Sucking Aged 3 to 6 Years
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ashraf, principal investigator, Cairo University
Other Study IDs: protocol89
Record Dates: First submitted 2016-10-15; First posted 2016-10-24 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Children With Digit Sucking

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine the prevalence of malocclusion among a group of Egyptian children with digit sucking aged 3 to 6 years.

DETAILED DESCRIPTION:
The purpose of the study is to determine the prevalence of malocclusion among a group of Egyptian children with digit sucking aged 3 to 6 years.

PICO:

Population: Egyptian Children with digit sucking aged 3 to 6 years. Outcome: Development of malocclusion.

ELIGIBILITY:
Inclusion Criteria:

* Children between ages 3 to 6 years.
* Children those are medically free.
* Both genders are included.
* Egyptian children

Exclusion Criteria:

* History of an obvious alternative cause for malocclusion (e.g. trauma, syndromes).
* Participants exposed to thumb sucking prevention programs.
* Participants who underwent orthodontic treatment for his/her malocclusion.
* Participants' caregivers refuse to give consent.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: population is limited to Egyptian children who are aged from 3 to 6 years and are thumb suckers. both genders are included
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Anterior open bite | 6 months
  Measured using a divider and the measurement is transferred onto a ruler. measuring unit is mm.
Over bite. | 6 months
  measured using a periodontal probe and the measurement is transferred onto a ruler. measuring unit mm.
Over jet. | 6 months
  measured using a periodontal probe and the measurement is transferred onto a ruler. measuring unit mm.
Anterior and posterior cross bite. | 6 months
  Observed visually.Binary units: (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hamdy, professor, Study Director — Cairo University; Salah Behery, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burford D, Noar JH. The causes, diagnosis and treatment of anterior open bite. Dent Update. 2003 Jun;30(5):235-41. doi: 10.12968/denu.2003.30.5.235. PMID 12861760
- [Background] Greenleaf S, Mink J. A retrospective study of the use of the Bluegrass appliance in the cessation of thumb habits. Pediatr Dent. 2003 Nov-Dec;25(6):587-90. PMID 14733476
- [Background] Kamdar RJ, Al-Shahrani I. Damaging oral habits. J Int Oral Health. 2015 Apr;7(4):85-7. PMID 25954079
- [Background] Larsson E. Sucking, chewing, and feeding habits and the development of crossbite: a longitudinal study of girls from birth to 3 years of age. Angle Orthod. 2001 Apr;71(2):116-9. doi: 10.1043/0003-3219(2001)0712.0.CO;2. PMID 11302587
- [Background] Moimaz SA, Garbin AJ, Lima AM, Lolli LF, Saliba O, Garbin CA. Longitudinal study of habits leading to malocclusion development in childhood. BMC Oral Health. 2014 Aug 4;14:96. doi: 10.1186/1472-6831-14-96. PMID 25091288
- [Background] Urzal V, Braga AC, Ferreira AP. Oral habits as risk factors for anterior open bite in the deciduous and mixed dentition - cross-sectional study. Eur J Paediatr Dent. 2013 Dec;14(4):299-302. PMID 24313582
- [Background] Warren JJ, Bishara SE. Duration of nutritive and nonnutritive sucking behaviors and their effects on the dental arches in the primary dentition. Am J Orthod Dentofacial Orthop. 2002 Apr;121(4):347-56. doi: 10.1067/mod.2002.121445. PMID 11997758
- [Background] Warren JJ, Levy SM, Nowak AJ, Tang S. Non-nutritive sucking behaviors in preschool children: a longitudinal study. Pediatr Dent. 2000 May-Jun;22(3):187-91. PMID 10846728
- [Background] Fisher, J.E.: Evidence-Based Psychotherapy. Springer, Reno, NV, 2006
- [Background] Ize-Iyamu IN, Isiekwe MC. Prevalence and factors associated with anterior open bite in 2 to 5 year old children in Benin city, Nigeria. Afr Health Sci. 2012 Dec;12(4):446-51. doi: 10.4314/ahs.v12i4.8. PMID 23513076
- [Background] Jajoo S et al. (2015). Oral Habits in School Going Children of Pune: A Prevalence Study. Journal of International Oral Health; 7(10):1-6.
- [Background] Jyoti S, Pavanalakshmi GP. Nutritive and Non-Nutritive Sucking Habits - Effect on the Developing Oro-Facial Complex; A Review. Dentistry 2014; 4(3)1-4.
- [Background] Katz CR, Rosenblatt A, Gondim PP. Nonnutritive sucking habits in Brazilian children: effects on deciduous dentition and relationship with facial morphology. Am J Orthod Dentofacial Orthop. 2004 Jul;126(1):53-7. doi: 10.1016/j.ajodo.2003.06.011. PMID 15224059
- [Background] Marwah N. Oral Habits. In: Text book of Pediatric Dentistry. 2nd ed. Jaypee Brothers Medical publishers; 2009. p. 281-298.
- [Background] W.H. Littlefield, B.D.S. (Durham), H.D.D. (Edinburgh). Thumb-sucking and its relationship to malocclusion in children. American Journal of Orthodontics, Volume 38, Issue 4, 293 - 300. 1952